CLINICAL TRIAL: NCT03484637
Title: Adherence to an Overweight and Obesity Treatment: the Evolution Chart
Brief Title: Response Evolution Chart
Status: Completed | Type: Observational
Sponsor: BiomediKcal (Other)
Responsible Party: Sponsor
Other Study IDs: BCE25318
Record Dates: First submitted 2018-03-25; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Obesity; Overweight; Motivation; Adherence, Patient
Keywords: motivation; Treatment adherence; Waist circumference; obesity; overweight
MeSH Terms: conditions — Obesity; Overweight; Patient Compliance; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lifestyle-medicine intervention: Photographic follow-up every 4 weeks
  Interventions: Other: Lifestyle-medicine intervention

INTERVENTIONS:
Other: Lifestyle-medicine intervention

SUMMARY:
This study evaluates patient response to a motivation evolution chart for a medical-nutrition intervention as a continuation of a previous study: adherence to an overweight and obesity treatment available at: https://www.ncbi.nlm.nih.gov/pubmed/25101227

ELIGIBILITY:
Inclusion Criteria:

* Voluntary assistance
* Clinical diagnosis of overweight
* Clinical diagnosis of obesity
* Patient desire to improve their aesthetic image and health status

Exclusion Criteria:

* This study does not consider patients who tried a diet to lose weight in the previous month or earlier

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Overweight and obese participants who consulted a medical nutrition clinic
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2018-03-24 (Actual)

PRIMARY OUTCOMES:
Evolution registration by photograph | 16 weeks
  To register Body Image of patients regarding results to a medical nutrition treatment

CONTACTS AND LOCATIONS:
Locations (1):
- BiomediKcal - Advanced Medical Nutrition & Lifestyle Center, Barranquilla, Atlántico, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuzmar IE, Cortes-Castell E, Rizo M. Effectiveness of telenutrition in a women's weight loss program. PeerJ. 2015 Feb 3;3:e748. doi: 10.7717/peerj.748. eCollection 2015. PMID 25674363
- [Background] Kuzmar I, Cortes E, Rizo M. Age group, menarche and regularity of menstrual cycles as efficiency predictors in the treatment of overweight. Nutr Hosp. 2014 Oct 30;31(2):637-41. doi: 10.3305/nh.2015.31.2.7501. PMID 25617544
- [Result] Kuzmar I, Rizo M, Cortes-Castell E. Adherence to an overweight and obesity treatment: how to motivate a patient? PeerJ. 2014 Jul 29;2:e495. doi: 10.7717/peerj.495. eCollection 2014. PMID 25101227